CLINICAL TRIAL: NCT02347033
Title: RCT of Sertraline Versus Cognitive Behavioural Therapy for Anxiety Symptoms in People With Generalised Anxiety Disorder Who Have Failed to Respond to Low Intensity Psychological Interventions as Defined by the NICE GAD Guidelines
Brief Title: Trial of Sertraline Versus Cognitive Behaviour Therapy for Generalised Anxiety
Acronym: ToSCA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties with recruitment during the internal pilot phase
Sponsor: University College, London (Other)
Collaborators: NHS Health Technology Assessment Programme (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/0249
Record Dates: First submitted 2015-01-16; First posted 2015-01-27 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Generalised Anxiety Disorder
Keywords: Sertraline; Selective Serotonin Reuptake Inhibitor (SSRI); Cognitive Behavioural Therapy (CBT); Increasing Access to Psychological Therapies (IAPT)
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Sertraline; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sertraline (Active Comparator): The pharmacological arm of the trial is the Selective Serotonin Reuptake Inhibitor (SSRI) Sertraline, prescribed at a daily dose of between 25 and 150mg by the patient's general practitioner (GP). If the medication is well tolerated and associated with reported clinical improvement we are asking the patients in this arm to continue taking it for 12 months.
  Interventions: Drug: Sertraline
- Cognitive Behavioural Therapy (CBT) (Active Comparator): The psychological therapy arm of the trial is Cognitive Behavioural Therapy (CBT) delivered by high intensity psychological therapists from local IAPT services. They will provide 14 to 16 sessions of a manualised treatment developed specifically for use in GAD and will be trained in its delivery.
  Interventions: Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Drug: Sertraline — Sertraline will be prescribed by the patients' GP, starting at 25mg daily for 1-2 weeks and increasing to 50mg daily if tolerated. The GP should review the patient within the first 2 weeks, checking for acceptability, concordance and any side-effects, with further reviews at 6 and 12 weeks. We expect the usual treatment dose to be 50 to 100mg daily, although some may require 150mg.
  We will suggest that the GPs use their usual procedures to review the patient's progress, asking about and noting functional change as well as clinical improvement. Minimal improvement after 12 weeks at a maximal tolerated dose should prompt consideration of change of treatment. If there has been an adequate therapeutic benefit there should be further review at 26 and 52 weeks.
  Other Names: SSRI
  Arms: Sertraline
Behavioral: Cognitive Behavioural Therapy — CBT will consist of 14 (+ / - 2) weekly 50-minute sessions and will cover 6 treatment modules: psychoeducation and worry awareness training; re-evaluation of the usefulness of worry; uncertainty recognition and behavioural exposure; problem-solving training; written exposure; and relapse prevention.
  Sessions will be digitally recorded and a random 10% assessed for quality (fidelity to the manual and therapist competence) by an independent external assessor according to pre-specified criteria. Patient consent for this will be obtained as part of obtaining informed consent.
  Other Names: CBT
  Arms: Cognitive Behavioural Therapy (CBT)

SUMMARY:
Generalised Anxiety Disorder (GAD) is common, causes unpleasant symptoms and impairs people's functioning. It is often chronic and may be accompanied by depression and other anxiety disorders. It is not currently clear whether medication or psychological therapy provides better long term outcomes for those not responding to simpler low intensity treatments so we propose to compare the clinical effectiveness of a pharmacological treatment (the drug Sertraline) with a Cognitive Behavioural Therapy (CBT) intervention.

Our hypothesis is that in people with GAD who have not responded to low intensity psychological interventions, CBT will lead to a greater improvement in their GAD symptoms as measured using the GAD-7 scale at 12 month follow-up than Sertraline.

DETAILED DESCRIPTION:
The investigators propose to undertake a randomised controlled trial (RCT) to compare the clinical effectiveness in terms of symptoms and function of a pharmacological treatment (the SSRI Sertraline) prescribed at therapeutic doses, with a manualised psychological intervention (Cognitive Behavioural Therapy, CBT) delivered by trained psychological therapists to patients with persistent generalised anxiety disorder (GAD) which has not improved with low intensity psychological interventions as defined by NICE (the National Institute for Clinical Effectiveness).

The investigators will recruit people via the Increasing Access to Psychological Therapies (IAPT) service from up to 15 sites in England. People still scoring highly on an anxiety measure (GAD-7) despite having received a low intensity psychological intervention will be given a brief flyer about the trial. Names of those interested in taking part who have given written consent to having their details released will be passed to the research team and the IAPT staff will also let the research team know the name of the participant's general practice, with their permission.

The research team will then contact potential participants offering them an appointment for an interview/assessment to discuss the study, sending them a patient information sheet to reach them at least 48 hours beforehand. The study information will explain that the medication being evaluated, Sertraline, although not currently licensed for GAD was recommended by NICE on the basis of its effectiveness in clinical trials and that the study team will be available to clarify any issues arising from this.

At the baseline assessment patients will be asked to give informed consent by a member of the research team and both medical suitability (as confirmed by fax/secure email from the GP) and the meeting of other inclusion/exclusion criteria will be checked. Upon confirmation of eligibility, baseline assessments will be carried out by a member of the research team and consenting patients randomised to receive either the medication or CBT. The Chief Investigator or other medically qualified persons within the research team will review all eligibility information and confirm that the patient is eligible.

Eligible participants will be randomised via an independent web-based computerised system to one of two interventions. The research team will provide the relevant contact details/instructions to patients in order to initiate treatment. The trial interventions consist of: (a) The medication sertraline prescribed by their GP according to a trial protocol matching current clinical recommendations and within a dosage between 25 and 150mg daily. We will ask GPs to review patients regularly (at least 6 times in 12 months) and patients to take the medication for a year unless they have significant adverse effects. Side-effects will be regularly monitored. (b) The other intervention is CBT delivered by high intensity therapists from local IAPT services. They will provide 14 to 16 sessions of a manualised treatment developed for use in GAD and will be trained in its delivery. The primary outcome will be the GAD-7 score measured at 12 months. Participants will also be asked to complete this outcome measure by postal questionnaire at 3, 6 and 9 months, as well as a range of secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Positive score of 10+ on GAD-7
* Primary diagnosis of GAD as diagnosed on MINI
* Failure to respond to NICE defined low intensity psychological interventions

Exclusion Criteria:

* Inability to complete questionnaires due to insufficient English or cognitive impairment;
* Current major depression
* Other comorbid anxiety disorder(s) of more severity or distress to the participant than their GAD;
* Significant dependence on alcohol or illicit drugs;
* Comorbid psychotic disorder, bipolar disorder;
* Treatment with antidepressants in past 8 weeks or any high intensity psychological therapy within past 6 months;
* Currently on contraindicated medication: monoamine oxidase Inhibitors within the past 14 days or pimozide;
* Patients with poorly controlled epilepsy;
* Known allergies to the Investigational Medicinal Product (IMP) or excipients;
* Concurrent enrolment in another Investigational Medicinal Product trial;
* Severe hepatic impairment;
* Women who are currently pregnant or planning pregnancy or lactating
* Patient on anti-coagulants
* History of bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
GAD-7 | GAD-7 score at 12 months
  A 7 item self-complete questionnaire with very good sensitivity (89%) and specificity (82%) for Generalised Anxiety Disorder (GAD).

SECONDARY OUTCOMES:
GAD-7 | GAD-7 score at 3 months
  A 7 item self-complete questionnaire with very good sensitivity (89%) and specificity (82%) for Generalised Anxiety Disorder (GAD).
GAD-7 | GAD-7 score at 6 months
  A 7 item self-complete questionnaire with very good sensitivity (89%) and specificity (82%) for Generalised Anxiety Disorder (GAD).
GAD-7 | GAD-7 score at 9 months
  A 7 item self-complete questionnaire with very good sensitivity (89%) and specificity (82%) for Generalised Anxiety Disorder (GAD).
HAM-A | HAM-A score at 12 months
  This is a 14 item observer rated anxiety scale which has been widely used, particularly in pharmacological studies widely used, particularly in pharmacological studies
Patient Health Questionnaire (PHQ-9) | PHQ-9 score at 3 months
  This is a 9 item self-rate scale widely used to monitor the severity of depression.
Patient Health Questionnaire (PHQ-9) | PHQ-9 score at 6 months
  This is a 9 item self-rate scale widely used to monitor the severity of depression.
Patient Health Questionnaire (PHQ-9) | PHQ-9 score at 9 months
  This is a 9 item self-rate scale widely used to monitor the severity of depression.
Patient Health Questionnaire (PHQ-9) | PHQ-9 score at 12 months
  This is a 9 item self-rate scale widely used to monitor the severity of depression.
Work and Social Activity Scale (WASAS) | WASAS score at 12 months
  This is a 5 item self-complete questionnaire which we will use to assess participants' difficulties with physical and social functioning
Euroquol-5 item-3 level (EQ-5D-3L) | Utility score at 3 months
  5 item, 3 level, self-completed measure of preference based generic health related quality of life. Utility scores calculated at each time point
Euroquol-5 item-3 level (EQ-5D-3L) | Utility score at 6 months
  5 item, 3 level, self-completed measure of preference based generic health related quality of life. Utility scores calculated at each time point scores for Quality Adjusted Life Years
Euroquol-5 item-3 level (EQ-5D-3L) | Utility score at 9 months
  5 item, 3 level, self-completed measure of preference based generic health related quality of life. Utility scores calculated at each time point scores for Quality Adjusted Life Years
Euroquol-5 item-3 level (EQ-5D-3L) | Utility score at 12 months
  5 item, 3 level, self-completed measure of preference based generic health related quality of life. Utility scores calculated at each time point scores for Quality Adjusted Life Years
Employment and Social Care Questionnaire (ESC) | ESC score at 6 months
  Relevant data on services used and productivity losses will be collected using this modified version of the Client Service Receipt Inventory
Employment and Social Care Questionnaire (ESC) | ESC score at 12 months
  Relevant data on services used and productivity losses will be collected using this modified version of the Client Service Receipt Inventory
(CSQ) Client Satisfaction Questionnaire | CSQ score at 3 months
  We are going to use the Client Satisfaction Questionnaire, a brief 8-item self-complete questionnaire as our treatment acceptability measure.
(CSQ) Client Satisfaction Questionnaire | CSQ score at 12 months
  We are going to use the Client Satisfaction Questionnaire, a brief 8-item self-complete questionnaire as our treatment acceptability measure.
Patient preference rating scale | Patient preference rating scale score at 12 months
  We are using a simple 4 item Likert scale used by our team in other studies

OTHER OUTCOMES:
Health service outcome - General practitioner (GP) contacts | GP contacts at 12 months
  We will collect relevant health service use data from both intervention arms at 12 months for the previous 12 months. This will include the number of GP contacts.
Health service outcome - Practice nurse contacts | Practice nurse contacts at 12 months
  We will collect relevant health service use data from both intervention arms at 12 months for the previous 12 months. This will include the number of practice nurse contacts.
Health service outcome - referrals to secondary care medical services | Referrals to secondary care medical services at 12 months
  We will collect relevant health service use data from both intervention arms at 12 months for the previous 12 months. This will include the number of referrals to secondary care medical services
Health service outcome - referrals to psychological therapy services | Referrals to psychological therapy services at 12 months
  We will collect relevant health service use data from both intervention arms at 12 months for the previous 12 months. This will include referrals to psychological therapy services.
Health service outcome - referrals to psychiatric services | Referrals to psychiatric services at 12 months
  We will collect relevant health service use data from both intervention arms at 12 months for the previous 12 months. This will include the number of referrals to psychiatric services.
Health service outcome - prescriptions for psychotropic medication | Prescriptions for psychotropic medication at 12 months
  We will collect relevant health service use data from both intervention arms at 12 months for the previous 12 months. This will include the number of prescriptions for psychotropic medication

CONTACTS AND LOCATIONS:
Overall Officials: Marta Buszewicz, Principal Investigator — University College, London
Locations (1):
- Camden & Islington (with Kingston), London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
To be discussed and decided by the Data Monitoring Committee